CLINICAL TRIAL: NCT00233077
Title: Patient Assistance to Reduce Breast Cancer Disparities
Brief Title: Patient Centered Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GCO 03-0593; 1R01CA10705-01A1 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Early-Stage Breast Cancer
Keywords: breast cancer; adjuvant treatment; racial disparities
MeSH Terms: conditions — Breast Neoplasms | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral: Patient Assistance (Experimental): Patient assistance programs
  Interventions: Behavioral: Patient Assistance
- Control: Information only (Other): Control patients will be sent a pamphlet about breast cancer & its treatment. We will call all patients 2 weeks later and ask if they received the packet. If they didn't, we will send the packet again.
  Interventions: Behavioral: Information only

INTERVENTIONS:
Behavioral: Patient Assistance — Patients will be surveyed to assess their knowledge about cancer & its treatment, experience with & access to health care system, trust, depression, social support & self-efficacy. A Brief Screening Needs Assessment will be done to ascertain practical, informational or psychosocial needs; based on their responses, an individualized action plan to connect with patient assistance programs will be created for the intervention group. We will ask intervention patients if they connected with any programs in their action plan. For those who didn't connect, we will give their name to an outreach worker. The outreach worker will call patients and identify reasons for not contacting the assistance programs.
  Arms: Behavioral: Patient Assistance
Behavioral: Information only — Control patients will be sent a pamphlet about breast cancer & its treatment. We will call all patients 2 weeks later and ask if they received the packet. If they didn't, we will send the packet again.
  Arms: Control: Information only

SUMMARY:
The purpose of this study is to determine whether patient-assistance programs as compared with usual care will help women with early stage breast cancer receive appropriate treatments.

DETAILED DESCRIPTION:
Numerous trials proved the efficacy of radiation following breast conserving surgery and systemic therapies to increase disease-free and overall survival among women with early-stage breast cancer. Yet 14%-89% of women do not receive them, especially minority women. Despite lower incidence of the disease, African American women are more likely than white women to die of breast cancer. As we near racial equity in rates of breast cancer screening, disparities in treatment and mortality remain. Efforts to achieve control of breast cancer and reduce racial disparities in mortality will not be fully realized until proven effective treatments are provided to those who can benefit.

Underuse of effective treatments may be caused by patient, physician and system factors. For breast cancer screening, women's lack of access to care; insurance; transportation; beliefs about fatalism and curability, and cancer's effect on partner relationships, all impact mammography rates. For breast cancer treatment, little is known about patient-related reasons for underuse, and less is known about racial differences in such reasons.

Interventions targeted to specific causes are more likely to succeed. For breast cancer screening, patient-centered interventions that successfully raise mammography rates among minority women include lay health workers to raise awareness about and address cultural beliefs and barriers to screening, vouchers to pay for screening and navigators to help women with abnormal screenings obtain needed follow-up. For breast cancer treatment, patient-assistance programs provide practical support such as financial counseling, aid with navigating the complex healthcare system, emotional support, and information about cancer and its treatment. Such programs abound but patients are often unaware of them. While these services may increase the receipt of effective adjuvant therapies, these strategies have not been rigorously tested.

We propose to conduct a randomized controlled trial to evaluate the effectiveness of patient-assistance programs as compared with usual care on receipt of adjuvant therapies among minority and nonminority women with newly operated early-stage breast cancer. During the 24 month trial, we will assess patients' beliefs about cancer and its treatment, and their practical, psychosocial, and informational needs and barriers to care. We will identify and train employees in existing cancer assistance services in order to increase the sustainability of this program beyond the grant-funded cycle. Specifically, we propose:

1. To assess racial differences in early-stage breast cancer patients' experiences, beliefs about and barriers to effective adjuvant treatments;
2. To evaluate the effectiveness of an intervention connecting women with early-stage breast cancer and cancer-related needs to community and hospital-based patient-assistance programs to reduce underuse of effective adjuvant breast cancer treatment overall and in minority populations and to assess its sustainability; and
3. To evaluate whether this patient assistance intervention affects patients' knowledge, attitudes and behaviors

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are English or Spanish speaking, with a new primary stage 1 or 2 breast cancer who have undergone either breast conserving surgery or mastectomy and those with tumors >1cm or <1cm and poorly differentiated;
* All surgeons performing breast surgery at the participating hospitals

Exclusion Criteria:

* Patients with dementia or those with a poor prognosis due to end-stage organ failure or other concomitant conditions such as those undergoing treatment for other cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
initiation and completion of primary treatment | Measured after completion of 6-mth interview

SECONDARY OUTCOMES:
adherence | Measured after completion of 6-mth interview
emotional and health status | Measured at baseline
emotional and health status | Measured after completion of 6-mth interview
patient satisfaction | measured at baseline
patient satisfaction | Measured after completion of 6-mth interview

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Bickell, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (8):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Metropolitan Hospital, New York, New York
  - Columbia University, New York, New York
  - Harlem Hospital Center, New York, New York
  - Albert Einstein College of Medicine, New York, New York
  - Montefiore Medical Center, New York, New York
  - Elmhurst Hospital Center, Queens, New York
  - Queens Hospital Center, Queens, New York

REFERENCES:
- [Derived] Guth AA, Fineberg S, Fei K, Franco R, Bickell NA. Utilization of Oncotype DX in an Inner City Population: Race or Place? Int J Breast Cancer. 2013;2013:653805. doi: 10.1155/2013/653805. Epub 2013 Dec 18. PMID 24455283
- [Derived] Bickell NA, Geduld AN, Joseph KA, Sparano JA, Kemeny MM, Oluwole S, Menes T, Srinivasan A, Franco R, Fei K, Leventhal H. Do community-based patient assistance programs affect the treatment and well-being of patients with breast cancer? J Oncol Pract. 2014 Jan;10(1):48-54. doi: 10.1200/JOP.2013.000920. Epub 2013 Sep 10. PMID 24023271
- [Derived] Lin JJ, Fei K, Franco R, Bickell NA. Breast cancer patients' recall of receiving patient assistance services. Springerplus. 2012 Oct 3;1:24. doi: 10.1186/2193-1801-1-24. eCollection 2012. PMID 23961354